CLINICAL TRIAL: NCT03262311
Title: Pimo Study: Extracellular Vesicle-based Liquid Biopsy to Detect Hypoxia in Tumours
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Institute of Cancer Research, United Kingdom (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: CCR4770
Record Dates: First submitted 2017-08-17; First posted 2017-08-25 (Actual); Last update posted 2019-12-23 (Actual); Status verified 2019-12

CONDITIONS: Cancer
MeSH Terms: conditions — Neoplasms | interventions — pimonidazole

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Hypoxia marker (Experimental): Administration of a single dose of the hypoxia marker Pimonidazole
  Interventions: Other: Hypoxia marker

INTERVENTIONS:
Other: Hypoxia marker — Single oral dose of pimonidazole 500 mg/m2
  Other Names: Pimonidazole

SUMMARY:
The purpose of this study is to test the potential of a relatively simple serum assay that aims to identify patient subpopulations whose curative radiotherapy outcome is likely to be compromised by radiobiological tumour hypoxia (prognostic value) and who are most likely to gain (predictive value) from the addition of radiation sensitiser drugs or targeted radiotherapy dose escalation.

DETAILED DESCRIPTION:
Aim: To analyse tiny cancer cell fragments called extracellular vesicles isolated from blood samples for their ability to identify patients with tumours that are relatively oxygen-starved and expected to be resistant to ionising radiation and many chemotherapy drugs.

Participants: 16 patients with proven cancer plus 4 healthy volunteers who give written informed consent to participate will be included in the study.

Recruitment: Eligible patients will be identified in the Outpatient Department at The Royal Marsden in Sutton or London and given a copy of the Information Sheet describing the study in detail. Dr Somaiah's team will call these potential volunteers at least 24 hours after they have received written information about the study to answer any questions. The same consent process will be followed for staff members who agree to participate as healthy volunteers. Research subjects who offer verbal agreement to participate will be asked for written consent and will be allocated a study ID. This will be used on all trial documentation and blood samples together with their initials and date of data/sample collection.

Pimonidazole administration: This well-established drug has the valuable property of binding exclusively to oxygen- starved tissues in a form that can be detected as a colour change in cell fragments released into the blood stream. A single oral dose of pimonidazole 500 mg/m2 will be prescribed and administered in a Royal Marsden outpatient clinic after confirmation of eligibility and completion of written informed consent. A member of the research team will monitor subjects to ensure that the prescribed drug is successfully taken (swallowed with water) before leaving the hospital (or going back to work/home in the case of healthy volunteers).

Blood sample: A peripheral venous blood sample of 20 ml will be collected from each participant the day after administration of pimonidazole, since it takes several hours for the drug to be absorbed and to bind to proteins and other molecules in oxygen-starved cells. A second sample will be collected 14 ±5 days later in order to confirm that all coloured cell fragments have disappeared from the circulation.

ELIGIBILITY:
Inclusion Criteria:

Patients i) Age ≥18 years ii) Biopsy-proven invasive carcinomas of head and neck, lung, bladder, uterine cervix or breast iii) Bulky (≥4 cm or ≥ 30 cc) primary/locally recurrent tumour or regional node masses iv) No clinical evidence of distant metastases unless oligometastases (ie distant relapse in only a limited number of regions for which local ablative therapy could be curative) v) Patient due for surgery, radiotherapy, systemic therapy or no anti-cancer treatment vi) Written informed consent

Healthy volunteers i) Age ≥18 years ii) Written informed consent

Exclusion Criteria:

Patients i) Inadequate cognitive ability to undertake the appropriate informed consent procedure

Healthy volunteers i) Past history of cancer, apart from non-melanomatous skin cancer or in situ carcinoma uterine cervix

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2017-11-10 (Actual); Primary Completion 2019-09-12 (Actual); Study Completion 2019-09-12 (Actual)

PRIMARY OUTCOMES:
Detectable pimonidazole staining | 24 hours and 2 weeks (+/- 5 days)
  Number of cancer patients with detectable pimonidazole staining in extracellular vesicles isolated from blood samples after a single dose of pimonidazole

CONTACTS AND LOCATIONS:
Overall Officials: Navita Somaiah, Principal Investigator — Institute of Cancer Research, United Kingdom
Locations (1):
- The Royal Marsden NHS Foundation Trust, Sutton, Surrey, United Kingdom